CLINICAL TRIAL: NCT00362791
Title: Multicenter Randomized Controlled Trial Evaluating the Efficacy of HIV/STD Prevention Counseling and Testing in Preventing High Risk Behaviors and New Sexually Transmitted Diseases (Project RESPECT)
Brief Title: Project RESPECT: The Efficacy of HIV/STD Prevention Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: San Francisco Department of Public Health (Other Government); City of Long Beach Department of Health and Human Services (Other Government); Colorado Department of Public Health and Environment (Other Government); Baltimore City Health Department (Other); City of Newark Health Department (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-1112.1; R30/CCR207113-03; R30/CCR307116-01; R30/CCR807114-04; R33/CCR907111-03; R30/CCR907117-03
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2006-08-10 (Estimated); Status verified 2005-07

CONDITIONS: HIV; Sexually Transmitted Diseases
Keywords: voluntary counseling and testing; HIV/STD prevention counseling; HIV/STD prevention intervention; counseling efficacy
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Health Belief Model

INTERVENTIONS:
Behavioral: "Enhanced HIV/STD Counseling:" 4 face-to-face, interctive counseling sessions based on the Theory of Reasoned Action & Health Belief Model
Behavioral: "Brief Counseling" (aka "client-centered counseling"): 2 brief, face-to-face interactive sessions targeted a patient-identified risk behavior
Behavioral: "HIV Prevention Education": 2 brief, didactic sessions informing the patient about HIV/STD prevention strategies

SUMMARY:
The efficacy of counseling to prevent infection with the human immunodeficiency virus (HIV) and other sexually transmitted diseases (STDs) has not been definitively shown. This multi-center randomized controlled trial (Project RESPECT) sought to compare the effects of 2 interactive HIV/STD counseling interventions with didactic prevention messages typical of current practice.

A total of 5758 STD clinic patients were enrolled from 5 public STD clinics (Baltimore, Md; Denver, Colo; Long Beach, Calif; Newark, NJ; and San Francisco, Calif) between July 1993 and September 1996. Eligible participants were heterosexual, HIV-negative patients aged 14 years or older who came for full STD examinations. Using a block design, participating men and women were randomzied separately to 1 of 3 individual face-to-face interventions. Arm 1 received "enhanced counseling" consisting of 4 interactive counseling sessions based on the Theory of Reasoned Action and Health Belief Model. Arm 2 received "brief counseling", consisting of 2 interactive risk-reduction sessions based on CDC's client-centered counseling model. Arms 3 and 4 each received 2 brief didactic messages about HIV/STD prevention messages typical of current care at that time. Participants assigned to Arms 1, 2, and 3 were actively followed up after enrollment with questionnaires at 3, 6, 9, and 12 months and STD laboratory examinations and tests at 6 and 12 months. An intent-to-treat analysis was used to compare interventions. Arm 4 participants were followed passively to determine potential effects of active study follow-up.

The main outcome measures were self-reported condom use and new diagnoses of STDs (gonorrhea, chlamydia, syphilis, HIV) defined by laboratory tests.

Results: At the 3- and 6-month follow-up visits, self-reported 100% condom use was higher (P<.05) in both the enhanced counseling and brief counseling arms compared with participants in the didactic messages arm. Through the 6-month interval, 30% fewer participants had new STDs in both the enhanced counseling (7.2%; P = .002) and brief counseling (7.3%;P=.005) arms compared with those in the didactic messages arm (10.4%). Through the 12-month study, 20% fewer participants in each counseling intervention had new STDs compared with those in the didactic messages arm (P = .008). Consistently at each of the 5 study sites, STD incidence was lower in the counseling intervention arms than in the didactic messages intervention arm. Reduction of STD was similar for men and women and greater for adolescents and persons with an STD diagnosed at enrollment.

Subset analyses found that

Based on these results, we conclude that short counseling interventions using personalized risk reduction plans can increase condom use and prevent new STDs. Effective counseling can be conducted even in busy public clinics.

DETAILED DESCRIPTION:
See Primary Paper:

Kamb ML, Fishbein M, Douglas, JM, Rhodes F, Rogers J, Bolan G, Zenilman J, Hoxworth T, Malotte CK, Iatesta M, Kent C, Lentz A, Graziano S, Byers RH, Peterman TA, Project RESPECT Study Group. Efficacy of risk reduction counseling to prevent human immunodeficiency virus and sexually transmitted diseases: a randomized controlled trial (Project RESPECT). JAMA 1998; 280:1161-1167

Also see:

Thompson DL, Douglas JM, Foster M, Hagensee ME, DiGuiseppi C, Barón AE, Cameron JE, Spencer TC, Zenilman J, Malotte CK, Bolan G, Kamb ML, Peterman TA for the Project RESPECT Study Group. HPV-16 Seroepidemiology in STD Clinics. J Infect Dis (in press).

Bolu OO, Lindsey C, Kamb ML, Kent C, Zenilman J, Douglas JM, Malotte CK, Rogers J, Peterman TA, for the Project RESPECT Study Group. Is HIV/STD Prevention Counseling Effective Among Vulnerable Populations? A Subset Analysis of Data Collected for a Randomized Controlled Trial Evaluating Counseling Efficacy (Project RESPECT) Sex Transm Dis 2004; 31(8): 469-74.

Gottlieb SL, Douglas JM, Foster M, Schmid DS, Newman DR, Baron AE, Bolan G, Iatesta M, Malotte CK, Zenilman J, Fisbhbein M, Peterman TA, Kamb ML, for the Project RESPECT STudy Group. Incidence of herpes simplex virus type 2 infection in five sexually transmitted disease clinics and the effect of HIV/STD risk reduction counseling. J Infect Dis 2004; 190: 1059-67.

Pealer Lisa, et al. Are Counselor Demographics Associated with Successful HIV/STD Prevention Counseling?" Sexually Transmitted Diseases (In press).

Warner L, Newman DR, Austin HA, Kamb ML, Douglas JM, Malotte CK, Zenilman JM, Rogers J, Bolan G, Fishbein M, Kleinbaum DG, Macaluso M, Peterman TA. Condom effectiveness for reducing transmission of gonorrhea and chlamydia: the importance of assessing partner infection status. Am J Epidemiol 2004; 159(3): 242-51.

Lyss SA, Kamb ML, Peterman TA, Moran JS, Newman DR, Bolan GA, Douglas JM, Jr., Iatesta M, Malotte CK, Zenilman J, Ehret J, Gaydos C, Newhall WJ, for the Project RESPECT Study Group. Chlamydia trachomatis among patients infected with and treated for Neisseria gonorrhoeae in sexually transmitted disease clinics in the United States. Annals Int Med, 2003; 139(3): 178-85.

Gottlieb SL, Douglas JM, Jr., Schmid DS, Bolan G, Iatesta M, Malotte CK, Zenilman J, Foster M, Baron AE, Steiner JF, Peterman TA, Kamb ML, for the Project RESPECT Study Group. Seroprevalence and correlates of herpes simplex virus type 2 infection in five Sexually Transmitted-Disease clinics. J Infect Dis 2002; 186 (15 November):

Fishbein M, Hennessy M, Kamb M, Bolan GA, Hoxworth T, Iatesta M, Fhodes F, Zenilman JM, for the Project RESPECT Study Group. Using intervention theory to model factors influencing behavior change: Project RESPECT. Evaluation and the Health Professions.2001; 4(24):363-384.

Lawrence JM, Zenilman J, Kamb ML, Iatesta M, Douglas JM, Rhodes F, Bolan G, Fishbein M, Peterman TA for the Project RESPECT Study Group. Sources of recent sexually transmitted disease (STD)-related health care for STD clinic patients. Sex Transm Dis 2001; 28(8): 1-4.

Diseker RA, Lin L, Kamb ML, Peterman TA, Kent C, Zenilman JM, Lentz A, Douglas JM, Rhodes F, Malotte CK, Iatesta M, for the Project RESPECT Study Group. Fleeting Foreskins: The misclassification of male circumcision status. Sex Transm Dis 2001; 28(6): 330-335.

Diseker RA III, Peterman TA, Kamb M, Kent C, Zenilman JM, Douglas JM, Rhodes F, Iatesta M. Circumcision and STD in the United States: cross-sectional and cohort analyses. Sex Transm Infect 2000; 76: 474-479.

Peterman TA, Lin LS, Newman DR, Kamb ML, Bolan G, Zenilman J, Douglas JM, Rogers J, Malotte CK, Project RESPECT Study Group. Does measured behavior reflect STD risk? Sex Transm Dis 2000; 27: 446-451.

Crosby R, Newman D, Kamb ML, Zenilman J, Douglas JM, Iatesta M, for the Project RESPECT Study Group. Misconceptions about STD protective behavior. Am J Prev Med 2000; 19 (3):167-173.

Malotte CK, Jarvis B, Fishbein M, Kamb ML, Iatatesta M, Hoxworth T, Zenilman J, Bolan G, for the Project RESPECT Study Group. Stage-of-change vs. an integrated psychosocial theory as a basis for developing effective behavior change interventions. AIDS Care 2000; 12:357-364.

Albarracin, D., Ho., R., McNatt, P. S., Williams, W. R., Rhodes, F., Malotte, C. K., Hoxworth, T., Bolan, G., Zenilman, J., Iatesta, M. & The Project RESPECT Study Group. Structure of beliefs about condom use. Health Psychology. 2000:19;458-468

Hennessy M, Bolan GA, Hoxworth T, Iatesta M, Rhodes F, Zenilman JM, Project RESPECT Study Group. Using growth curves to determine the timing of booster sessions. Structural Equation Modeling 1999; 6(4): 322-342.

Kamb ML, Rhodes F, Hoxworth T, Rogers J, Lentz A, Kent C, Peterman TA, MacGowan R, Project RESPECT Study Group. What about money? Effect of small monetary incentives on enrollment, retention, and motivation to change behavior in an HIV/STD prevention counseling intervention. Sex Transm Infect 1998; 74:253-255.

McGill W, Miller K, Bolan G, Malotte K, Zenilman J, Iatesta M, Kamb ML, Douglas JM, Jr. for the Project RESPECT Study Group. Awareness of and experience with the female condom among patients attending STD clinics. Sex Transm Dis 1998; 25(4): 222-223.

ELIGIBILITY:
Inclusion Criteria:

- patients who came to the STD clinic and who were eligible in routine clinic practice to undergo confidential HIV testing

Exclusion Criteria:

* residence outside the clinics' catchment areas
* had made firm plans (e.g., can give a new address) to move outside the clinic catchment area during the next 12 months
* unable to provide informed consent to be tested for HIV and take part in the follow up aspect of the study (e.g., incarcerated, mental status changes from drugs, alcohol, medication)
* reported that he or she had tested positive for HIV in the past
* did not speak and comprehend English well enough to participate in the interventions
* came to the clinic for something other than a full routine STD clinic examinations
* was a man who reported sex with a man in the past 12 months
* had been approached for study participation on a previous clinic visit, and hd already enrolled or refused participation
* age < 14 years.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000
Dates: Start 2003-04; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Kamb, MD, MPH, Principal Investigator — US Centers for Disease Control and Prevention (CDC)